CLINICAL TRIAL: NCT04222491
Title: Outcomes of Clinical Food Oral Immunotherapy for Peanut Allergy
Brief Title: Food Oral Immunotherapy for Peanut Allergy
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003564
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Peanut Allergy
Keywords: food allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This is an open label observational single center study of clinical food oral immunotherapy outcomes with biomarker samples and participant and/or caregiver-completed questionnaires in participants between 6 months and 65 years of age with IgE-mediated peanut allergy undergoing food oral immunotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- active peanut OIT (Experimental): active peanut oral immunotherapy
  Interventions: Drug: Peanut oral immunotherapy

INTERVENTIONS:
Drug: Peanut oral immunotherapy — Peanut oral immunotherapy for peanut allergy
  Other Names: Peanut flour; Peanut allergen powder

SUMMARY:
This is an open label observational single center study of clinical food oral immunotherapy outcomes with biomarker samples and participant and/or caregiver-completed questionnaires in participants between 6 months and 65 years of age with IgE-mediated peanut allergy undergoing food oral immunotherapy.

DETAILED DESCRIPTION:
In this research study the investigators want to learn more about the experience of participants with peanut allergy and their caregivers undergoing food oral immunotherapy (OIT) for peanut allergy. Food oral immunotherapy (OIT) is a treatment for individuals with a food allergy to reduce the body's allergic response to the food allergen, resulting in fewer symptoms. The treatment is also called desensitization. An individual becomes desensitized to the food allergen by ingesting small amounts of the food that are slowly increased. Over time, this helps the body's immune system become used to the food so that it no longer causes an allergic reaction. By desensitizing to peanut, it may lower the risk of life-threatening allergic reactions and cause a decreased sensitivity to peanut. The investigators specifically want to learn more about the effects of food OIT on quality of life and other outcomes important to participants with peanut allergy and their caregivers and to ultimately develop tests to predict who may respond favorably to food OIT.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 6 months and 65 years of age with a diagnosis of immunoglobulin E (IgE)-mediated peanut allergy and their caregivers; a diagnosis of IgE-mediated peanut allergy is defined by: (1) documented history of peanut allergy or determined to be allergic by oral food challenge; (2) evidence of peanut-specific IgE by either: positive skin prick test to peanut allergen (reaction wheal at least 3 mm larger than saline control) or serum peanut-specific IgE > 0.34 kilo-unit/liter (kU/L) or international unit/milliliter (IU/mL) at screening visit
* Referral by Massachusetts General Hospital (MGH) allergist for food oral immunotherapy
* Willing to sign informed consent or whose caregiver is willing to sign the informed consent (age appropriate)
* Willing to sign the assent form, if age appropriate

Exclusion Criteria:

* History of severe or life-threatening episode of anaphylaxis or anaphylactic shock within 60 days of screening
* Severe or poorly controlled asthma
* Diagnosis of other severe or complicating medical problems, including autoimmune or chronic immune inflammatory conditions or gastrointestinal inflammatory conditions, such as inflammatory bowel diseases and eosinophilic gastrointestinal disorders
* Current use of beta blocker medication(s)
* Inability to cooperate with and/or perform oral food challenge procedures
* Females who are pregnant, planning to become pregnant, or breastfeeding
* Investigator determination of safety concern for any reason

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who tolerate the maintenance dose of 300 mg peanut protein with no symptoms within two years of starting OIT | 2 years
  Feasibility analysis as assessed by the proportion of participants who tolerate the maintenance dose in a dichotomous manner

SECONDARY OUTCOMES:
Change in quality of life scores from baseline to end of treatment | 4 years
  Change in quality of life scores from baseline assessment to end of treatment assessment using the Food Allergy Quality of Life Questionnaire (FAQLQ) total score. The FAQLQ total and domain scores range from 1-7 where 1 was the best possible score (i.e. fewest problems or better health related quality of life) and with the total score being the average of the domain scores. The domains include Emotional Impact, Social and Dietary Restrictions, and Food Anxiety.
Change in peanut specific serum immunoglobulin E (IgE) from baseline to end of treatment | 4 years
  Change in peanut specific serum immunoglobulin E (IgE) [in kilo-units per liter (kU/L) or international units per milliliter (IU/mL)] from baseline to end of treatment
Change in skin prick test reactivity to peanut extract from baseline to end of treatment | 4 years
  Change in skin prick test wheal diameter measurement in millimeters to peanut extract from baseline to end of treatment
The proportion of participants who tolerate a cumulative dose of 5000 mg peanut protein on oral food challenge without treatment after 12 months on maintenance dose | 4 years
  Desensitization to peanut as assessed by cumulative tolerated dose
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 4 years
  Safety analysis as assessed by patient-reported or observed allergic symptoms that will be analyzed and tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No